CLINICAL TRIAL: NCT06931158
Title: Optimizing Open Placebos for Chronic Pain Patients
Brief Title: HOnest Placebos With Explanations: Evaluating Open-Label Placebos for Chronic Pain
Acronym: HOPE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rhode Island Hospital (Other)
Responsible Party: Principal Investigator, Michael Bernstein, Assistant Professor, Rhode Island Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RIH-2053624-7
Record Dates: First submitted 2025-04-01; First posted 2025-04-17 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Chronic Low-back Pain; Chronic Pain
Keywords: open-label placebo; rationales; placebo effect
MeSH Terms: conditions — Chronic Pain | interventions — Mindfulness

STUDY DESIGN:
Masking Description: Participants are blind to the research hypothesis but not to treatment allocation that are by definition open.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- OLP + Standard Rationale (Experimental): Participants in this group will receive an open-label placebo along with information based on the standard rationales used in other OLP studies.
  Interventions: Drug: Open-label Placebo; Behavioral: Standard Rationale
- OLP + Mindfulness Rationale (Experimental): Participants in this group will receive an open-label placebo along with information with mindfulness information.
  Interventions: Drug: Open-label Placebo; Behavioral: Mindfulness
- OLP + Control Rationale (Placebo Comparator): Participants in this group will receive an open-label placebo along with no information on the placebo effect.. They will receive basic epidemiological information on chronic pain to guarantee structural equivalence of the trial design.
  Interventions: Drug: Open-label Placebo; Behavioral: Control Rationale
- No Treatment + Control Rationale (Sham Comparator): Participants in this group will receive no treatment. They will receive basic epidemiological information on chronic pain to guarantee structural equivalence of the trial design.
  Interventions: Behavioral: Control Rationale

INTERVENTIONS:
Drug: Open-label Placebo — Open-label placebo pill for 21 days at 2 per day
  Other Names: OLP; Zeebo
  Arms: OLP + Control Rationale; OLP + Mindfulness Rationale; OLP + Standard Rationale
Behavioral: Standard Rationale — Scientific rationale about the placebo effect
  Arms: OLP + Standard Rationale
Behavioral: Mindfulness — Mindfulness based rationale
  Arms: OLP + Mindfulness Rationale
Behavioral: Control Rationale — Basic epidemiological information about chronic pain to achieve structural equivalence for the control groups
  Arms: No Treatment + Control Rationale; OLP + Control Rationale

SUMMARY:
The goal of this clinical trial is to examine the effect of rationale condition when taking open-label placebos on pain by 1) comparing each rationale to the no rationale control condition and the no treatment control condition; and 2) comparing the rationale conditions to each other. We also aim to examine the effect of rationale condition on prescription opioid use by 1) comparing each rationale to the no rationale control condition and the no treatment control condition; and 2) comparing the rationale conditions to each other.

This study will include patients with chronic low back pain. The main question it aims to answer is:

How do rationales influence the effects of open-label placebos?

Researchers will compare different rationales given when taking an open-label placebo and a no-treatment group and a no rationale group taking OLPs.

ELIGIBILITY:
Inclusion criteria are:

* chronic pain (pain lasting at least 3 months, pain intensity 4/10 or over and interference 3/10 or over)
* at least 18 years old
* English speaking
* have a smartphone or computer with video access
* the chronic pain is concentrated into the patient's lower back (tentative criteria based on recruitment rate)

Exclusion Criteria

* Have chronic pain because of a cancer diagnosis
* Over 89 years of age
* Suspect an allergy to any placebo ingredient
* Currently receiving worker's compensation.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 340 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Pain intensity | across 42 days
  Single-item assessing current pain level from 0 (min value) to 10 (max value). Higher scores indicate more pain intensity

SECONDARY OUTCOMES:
Pain interference | across 42 days
  Pain Interference subscale from Brief Pain Inventory Pain interference is measured for general activity, mood, walking ability, work, relationships, sleep, and enjoyment of life on a 0-10 NRS with 0 = "does not interfere" and 10 = "completely interferes" Higher scores indicated greater pain intensity or greater interference with function.
Pain catastrophizing | across 42 days
  Single item assessing how much the patient catastrophizes about their pain from 0 (minimum) to 10 (maximum). Higher scores indicate more catastrophizing.
  13 items rated on 5-point Likert scales, from (0) not at all to (4) all the time Higher score indicates higher level of catastrophizing
  Item scores are summed into a total score (PCS-T) and three subscale scores:
  * Rumination (PCS-R): Items 8, 9, 10, and 11
  * Magnification (PCS-M): Items 6, 7, 13
  * Helplessness (PCS-H): Items 1, 2, 3, 4, 5, and 12 Minimum total score = 0, maximum total score = 52 Subscale score ranges: PCS-R: 0-16; PCS-M: 0-12; PCS-H: 0-24 A total score above 30 indicates clinically relevant level of catastrophizing
Prescription Medication use (including opioids) | across 42 days

OTHER OUTCOMES:
Placebo use | across 21 days

CONTACTS AND LOCATIONS:
Locations (1):
- Rhode Island Hospital, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: Undecided